CLINICAL TRIAL: NCT00489424
Title: A Randomized, Multicenter, Double-blind, Double-dummy, Parallel-group Study of Acetaminophen or Fluvastatin Compared to Placebo on the Transient Post-Dose Symptoms (PDS) Following an i.v. Infusion of a Single Dose of Zoledronic Acid 5mg, in Post-menopausal Women With Low Bone Mass
Brief Title: Acetaminophen or Fluvastatin Compared to Placebo on the Transient Post-Dose Symptoms (PDS) Following an Intravenous (i.v.) Infusion of a Single Dose of Zoledronic Acid 5mg, in Post-menopausal Women With Low Bone Mass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446HUS136
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2009-09-14 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Osteoporosis
Keywords: zoledronic acid; post dose symptoms; transient; acetaminophen; fluvastatin
MeSH Terms: conditions — Osteoporosis | interventions — Acetaminophen; Fluvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Acetaminophen (Experimental): 2 capsules of acetaminophen 325 mg and 2 capsules of placebo (matching fluvastatin) administered 45 +/- 15 minutes prior to i.v. infusion of zoledronic acid 5 mg, then 2 capsules of acetaminophen 325 mg 4 times per day (including medication taken at study site at visit 2/day 1) over the next 3 days (not exceeding 8 capsules in a 24-hour period).
  Interventions: Drug: Acetaminophen
- Fluvastatin (Experimental): 2 capsules of fluvastatin 40 mg and 2 capsules of placebo (matching acetaminophen) administered 45 +/- 15 minutes prior to i.v. infusion of zoledronic acid 5 mg, then 2 capsules of placebo (matching acetaminophen) 4 times per day (including medication taken at study site at visit 2/day 1) over the next 3 days (not exceeding 8 capsules in a 24-hour period).
  Interventions: Drug: Fluvastatin
- Placebo (Placebo Comparator): 2 capsules of placebo (matching fluvastatin) and 2 capsules of placebo (matching acetaminophen) administered 45 +/- 15 minutes prior to intravenous (i.v.) infusion of zoledronic acid 5 mg, then 2 capsules of placebo (matching acetaminophen) 4 times per day (including medication taken at study site at visit 2/day 1) over the next 3 days (not exceeding 8 capsules in a 24-hour period).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Acetaminophen
  Arms: Acetaminophen
Drug: Fluvastatin
  Arms: Fluvastatin

SUMMARY:
This study will evaluate the efficacy of acetaminophen or fluvastatin in reducing the rate of occurrence and the severity of post dose symptoms that may occur during the 3 day period following a zoledronic acid infusion in post menopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women greater than or equal to 45 and less than or equal to 79 years of age at randomization
2. Women who are clinically indicated for treatment with Bisphosphonates for osteopenia or osteoporosis with a documented central (spine or hip) Bone Mineral Density T Score less than or equal to 1.5

Exclusion Criteria:

1. Any prior treatment with intravenous Bisphosphonates
2. Oral treatment with Bisphosphonates for more than 8 weeks or within 6 months prior to the screening visit
3. Patients who are taking, and are unwilling or unable to stop taking, certain medications
4. Patients who require anticoagulant therapy
5. Patients with a known hypersensitivity to ibuprofen, ACET, bisphosphonates, statins or with allergies manifested by attacks of asthma, urticaria or acute rhinitis following
6. Proteinuria (protein detected on a urine dipstick) greater than or equal to 2+ at screening
7. Protocol specific laboratory values that fall out of range for this study
8. Ongoing infection (oral body temperature greater than or equal to 37.5C (99.5°F),chronic febrile disease or fever of unknown origin at screening or randomization
9. Active dental infection, unhealed dental extraction or planned oral surgery within 3 months after randomization
10. History of iritis, uveitis or chronic conjunctivitis
11. History of hypoparathyroidism, hyperparathyroidism or Paget's Disease
12. Partial or total removal of parathyroid or thyroid gland
13. History of malignancy of any organ system, treated or untreated, within the past 1 year whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
14. Treatment with an investigational drug within the previous 30 days of screening
15. Patients with any medical or psychiatric condition which, in the opinion of the Principal Investigator, would preclude the participant from adhering to the protocol or completing the trial per protocol, or any patient who the Principal Investigator thinks should not participate in the study for any reason, including current drug or alcohol abuse

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 45 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Refer to the E-portal link for ZOL446HUS136, Http://www.osteoporosisclinicalresearch.com, New Jersey, United States

REFERENCES:
- See also: Click here for more information on this study — http://www.osteoporosisclinicalresearch.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Started | 267 | 264 | 262
Completed | 263 | 259 | 257
Not Completed | 4 | 5 | 5
Not completed — Adverse Event | 3 | 3 | 4
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Administrative problems | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acetaminophen | Fluvastatin | Total
Number analyzed (Participants) | 267 | 264 | 262 | 793
Age, Customized [Number; unit: participants]
  Between 45 and 55 years | 64 | 69 | 67 | 200
  Between 56 and 64 years | 102 | 98 | 92 | 292
  >=65 years | 101 | 97 | 103 | 301
Sex/Gender, Customized [Number; unit: participants]
  Female | 267 | 264 | 262 | 793

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Clinically Significant Increase in Oral Body Temperature or Use of Rescue Medication.
Description: Clinically significant increase in oral body temperature or used rescue medication ibuprofen >= 1 time during the 3-day period after i.v. infusion of zoledronic acid 5 mg. A clinically significant increase in body temperature was defined as an increase of at least 1 degree Celsius from baseline and a mean oral body temperature reading of at least 38.5 degrees Celsius occurring at least once during the 3-day treatment period.
Time Frame: 0 - 3 days
Population: Intent to Treat (ITT) population.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 267 | 264 | 262
proportion of patients
  Increase in oral body temperature:Yes | 0.607 | 0.398 | 0.618
  Increase in oral body temperature:No | 0.39 | 0.602 | 0.382

2. Secondary Outcome: Proportion of Patients With a Clinically Significant Increase in Oral Body Temperature.
Description: Clinically significant increase in oral body temperature >= 1 time during the 3-day period after i.v. infusion of zoledronic acid 5 mg. A clinically significant increase in body temperature was defined as an increase of at least 1 degree Celsius from baseline and a mean oral body temperature reading of at least 38.5 degrees Celsius occurring at least once during the 3-day treatment period.
Time Frame: 0 - 3 days
Population: Intent to Treat (ITT) population.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 267 | 264 | 262
proportion of patients
  Increase in oral body temperature: Yes | 0.105 | 0.049 | 0.115
  Increase in oral body temperature: No | 0.891 | 0.951 | 0.885

3. Secondary Outcome: Proportion of Patients Who Used Rescue Medication.
Description: Patients that took rescue medication >= 1 time during the 3-day period after i.v. infusion of zoledronic acid 5 mg. Patients who experienced severe discomfort after their first home measurements and self-administration of study medication were allowed to take ibuprofen (200 mg tablets every 4-6 hours as needed) as rescue medication while continuing to take their study medication.
Time Frame: 0 - 3 days
Population: Intent to Treat (ITT) population. One patient who used rescue medication in acetaminophen arm and two patients in fluvastatin arm were not included in analysis due to lack of documentation regarding use and exposure of rescue medication.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 267 | 264 | 262
proportion of patients
  Took rescue medication >= 1 time: Yes | 0.573 | 0.386 | 0.595
  Took rescue medication >= 1 time: No | 0.423 | 0.614 | 0.405

4. Secondary Outcome: Number of Rescue Medication Tablets Taken
Description: Patients who experienced severe discomfort after their first home measurements and self-administration of study medication were allowed to take ibuprofen (200 mg tablets every 4-6 hours as needed) as rescue medication while continuing to take their study medication.
Time Frame: 0 - 3 days
Population: Number of patients who took rescue medication at least once. One patient in acetaminophen arm was not included in analysis since the number of tablets taken was not recorded.
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 153 | 102 | 158
tablets | 6.3 (4.41) | 5.7 (4.73) | 6.5 (4.78)

5. Secondary Outcome: Time to First Rescue Medication After Infusion of Zoledronic Acid 5 mg.
Description: as for outcome 4
Time Frame: 0 - 3 days
Population: Number of patients who took rescue medication at least once. Two patients who took rescue medication in fluvastatin arm were not included in analysis since the time rescue medication was taken was not recorded.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 153 | 103 | 156
hours | 21.9 (12.21) | 28.2 (18.15) | 19.9 (40.95)

6. Secondary Outcome: Proportion of Patients With a Major Increase (Worsening) in Severity of Questionnaire Symptoms.
Description: A major increase (worsening) in severity was defined as an increase in severity of 2 units or more from baseline at least once during the 3 days immediately following i.v. infusion of zoledronic acid 5 mg. The severity of the symptom was evaluated using a 4-point categorical scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: 0 - 3 days
Population: Intent to Treat (ITT) population.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 267 | 264 | 262
proportion of patients
  Feeling feverish | 0.395 | 0.235 | 0.397
  Headache | 0.391 | 0.254 | 0.439
  Aches and pains of muscles/joints | 0.477 | 0.337 | 0.462

7. Secondary Outcome: Proportion of Patients Reporting Severe Questionnaire Symptoms.
Description: A severe questionnaire symptom was defined as experiencing a severe specified symptom (feeling feverish, experiencing headaches, having aches and pains of muscles and joints) at least once post-baseline.
Time Frame: 0 - 3 days
Population: Intent to Treat (ITT) population.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 267 | 264 | 262
proportion of patients
  Feeling feverish | 0.135 | 0.076 | 0.145
  Headache | 0.157 | 0.068 | 0.160
  Aches and pains of muscles/joints | 0.303 | 0.212 | 0.302

8. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Measurement of Symptom Severity
Description: Effect on severity of symptoms following i.v. infusion of zoledronic acid 5 mg. The VAS is a 100-mm linear visual analog scale (0 = no symptoms to 100 = severe symptoms). The baseline VAS measurement was defined as the VAS measurement recorded prior to the infusion.
Time Frame: 0 - 3 days
Population: Intent to Treat (ITT) population. Number of participants analyzed may vary from ITT population due to some patients not reporting baseline or post baseline VAS measurement. Calculating change requires both baseline and post baseline values to be present.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Number analyzed (Participants) | 267 | 264 | 262
units on a scale
  Change from baseline to Day 1 - late evening | 7.6 (22.74) | 4.4 (18.00) | 6.0 (18.89)
  Change from baseline to Day 2 - late evening | 18.9 (25.86) | 11.8 (23.22) | 20.8 (27.18)
  Change from baseline to Day 3 - late evening | 6.2 (19.66) | 3.9 (17.59) | 6.6 (20.40)

ADVERSE EVENTS:
Time Frame: At the end of study
Description: Safety Population
Arm/Group | Placebo | Acetaminophen | Fluvastatin
Serious Adverse Events (participants affected / at risk) | 1/267 | 2/264 | 2/262
Other Adverse Events (participants affected / at risk) | 34/267 | 39/264 | 36/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=267) | Acetaminophen (N=264) | Fluvastatin (N=262)
Uveitis (Eye disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=267) | Acetaminophen (N=264) | Fluvastatin (N=262)
Nausea (Gastrointestinal disorders) | 7 | 16 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 9 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 11 | 10
Headache (Nervous system disorders) | 8 | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.